CLINICAL TRIAL: NCT05637333
Title: Study Examining if Sonazoid is an Effective Contrast Agent to Identify Myocardial Perfusion
Brief Title: Sonazoid in Myocardial Perfusion Imaging
Acronym: (SIMPI)
Status: Withdrawn | Type: Observational
Why Stopped: Study classed as CTIMP
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRC/2022/004
Record Dates: First submitted 2022-10-12; First posted 2022-12-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Diagnostic Imaging; Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Contrast Stress Echocardiography — Dipyridamole will be infused at 0.56mg/kg of body weight over 4mins. After 2 minutes, if the patient has tolerated the infusion well, a further 0.28mg/kg will be infused over 2 minutes. Tolerance will be determined by the absence of 1) myocardial ischaemia (significant chest pain with ECG ST depression or T wave inversion or wall motion abnormality on ECHO) 2) a significant drop in blood pressure 3) significant arrhythmia and 4) intolerable symptoms. One minute after completion of Dipyridamole infusion Sonazoid will be infused at the same rate as was used during acquisition of the rest images. After 45 seconds when steady state is reached, the ultrasound images will be acquired as stated below in contrast imaging. If the Dipyridamole is not well tolerated by one minute after the 0.56mg/kg infusion, we will move straight to the infusion of Sonazoid with no extra 0.28mg/kg infusion.

SUMMARY:
Currently, Sonazoid is mainly used for imaging liver lesions by assessing perfusion characteristics. However, the ultrasound technology is the same as for cardiac imaging and the stability of the microbubbles will potentially aid the detection of myocardial perfusion defects. This study will look at the feasibility of using sonozoid in this way.

DETAILED DESCRIPTION:
Ultrasound contrast agents are gas-filled microbubbles that enhance the visualisation of cardiac structures, function and blood flow. Myocardial contrast echocardiography enables us to visualise myocardial perfusion and provides incremental information for diagnosis of coronary artery disease (CAD) and prognosis beyond wall motion assessment .

Using ultrasound at low acoustic power (low/intermediate MI) causes the microbubbles to oscillate resulting in giving off non-linear signals which are different from tissues which gives off linear signals.

The first contrast agents were used in 1968. Since then the technology has been refined and now the microbubbles are more stable and consist of an inert gas encapsulated in a lipid or albumin shell. These microbubbles remain intact in the systemic circulation because of their small size can transit through the pulmonary circulation.

The indication for myocardial perfusion imaging is when vasodilator stress like Dipyridamole is performed. Vasodilators do not readily induce wall motion abnormalities but cause perfusion defects to occur which allows detection of CAD. Myocardial perfusion imaging is also indicated during treadmill or dobutamine stress when suspicion of CAD is high as it is more sensitive than wall motion for the detection of CAD.

Myocardial perfusion imaging looks at a uniformity of contrast appearance in the myocardium, following a continuous microbubble infusion. If there is decreased perfusion, the appearance of contrast will be delayed and the opacification will not be uniform.

The advantage of Sonazoid over the other frequently used contrast agents (Sonovue, Luminity, Optison) is that the microbubbles are more robust, allowing for a higher MI setting to be used during scanning. The higher MI setting enhances higher intensity bubble signal with improved spatial and temporal resolution which improves image quality and diagnostic accuracy.

This study is not looking for diagnosis in patients, which will be done according to standard of care. It is to evaluate whether it is possible to assess myocardial perfusion using the contrast agent Sonazoid.

ELIGIBILITY:
Inclusion Criteria:

* Positive and normal Clinical SE
* Able to provide informed consent

Exclusion Criteria:

* Unable / unwilling to give informed consent
* Allergy to Perfluorobutane
* Egg allergy
* Patients with right to left arteriovenous cardiac or pulmonary shunt
* Unstable heart disease
* Serious pulmonary disease
* Pregnancy or lactation Women of child bearing potential (defined as not chemically or surgically sterilised or post menopausal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients will be identified for this proof of concept study.
  Patients who have already had a positive clinical stress echo scan will be approached about participating in this study
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
To demonstrate if sonazoid gives adequate opacification of the myocardium at low mechanical index using stress echocardiography | 1 day
  Contrast Stress echocardiography (SE) using sonazoid will be used to predict if patients with very low probability of CAD have flow-limiting coronary stenosis>70% in any major coronary artery branches in patients with previous significant (>2 contiguous segments) inducible ischemia on stress echocardiography (SE).
To demonstrate if sonazoid gives adequate opacification of the myocardium at intermediate mechanical index using stress echocardiography | 1 day
  Contrast Stress echocardiography (SE) using sonazoid will be used to predict if patients with very low probability of CAD have flow-limiting coronary stenosis>70% in any major coronary artery branches in patients with previous significant (>2 contiguous segments) inducible ischemia on stress echocardiography (SE).

SECONDARY OUTCOMES:
Myocardial blood flow reserve assessment for prediction of flow-limiting CAD | 1 day
  Myocardial blood flow will be measured during the scan

CONTACTS AND LOCATIONS:
Overall Officials: Roxy Senior, MD, Principal Investigator — LNWUH NHS Trust
Locations (1):
- London North West University Healthcare NHS Trust, Harrow, Middx, United Kingdom

IPD SHARING:
Plan to Share IPD: No